CLINICAL TRIAL: NCT00588419
Title: Quantification of Breast Sensation Following Postmastectomy Breast Reconstruction
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 06-047
Record Dates: First submitted 2007-12-24; First posted 2008-01-08 (Estimated); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Breast Cancer; Cancer
Keywords: Breast Cancer; Cancer; Breast Sensation; Postmastectomy Breast Reconstruction
MeSH Terms: conditions — Breast Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- 1: Patients who have undergone mastectomy Patients who have undergone immediate, twostage expander/implant breast reconstruction; Patients who have undergone immediate, autogenous tissue flap reconstruction including: pedicled and/or free TRAM flap or DIEP flap reconstruction
  Interventions: Behavioral: breast exam and questionaire

INTERVENTIONS:
Behavioral: breast exam and questionaire — A physical examination of your breast(s), we will ask you to complete a short questionnaire that asks questions regarding sensations in your reconstructed breast(s) and another short questionnaire that asks questions regarding your medical and surgical history. The physical examination and the questionnaires will be completed in the outpatient clinic. This should take about 30 minutes to complete.

SUMMARY:
The purpose of this study is to evaluate the return of sensation in the breast(s) following breast mastectomy with and without reconstruction. Four different sensations: touch, vibration, superficial pain, and temperature will be evaluated. In addition, we will look at factors that may contribute to the return of breast sensations.

DETAILED DESCRIPTION:
This study entitled "The Quantification of Breast Sensations Following Postmastectomy Breast Reconstruction" will evaluate the recovery of sensation in the reconstructed as well as in the nonreconstructed breast. Touch, vibration, pain and temperature sensation will be objectively evaluated greater than 1 year following completion of reconstruction. Breast sensation following immediate, tissue expander/implant breast reconstruction will be compared with that following immediate, autogenous tissue reconstruction.

A formal sensory examination will be performed. SemmesWeinstein monofilaments will evaluate touchpressure sensation in the breast. A Bioesthesiometer will determine the recovery of vibratory sensation. Temperature sensation will be evaluated by application of warm and cool stimuli. Superficial pain sensation will be evaluated by application of sharp and dull stimuli.

A patient reported assessment of sensory changes in the breast will be administered to patients. The Breast Sensation Assessment Scale © is designed to measure the prevalence, severity, and distress of 18 different sensory symptoms following breast surgery. A "Patient Demographic and Treatment Information Form" and patients' medical records will be used to obtain demographic and treatment data. The role of confounding variables (including: patient age, breast volume, axillary procedures performed and adjuvant therapies received) on the recovery of sensation will be evaluated.

The estimated accrual time for this study is 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone mastectomy
* Patients who have undergone immediate, twostage expander/implant breast reconstruction
* Patients who have undergone immediate, autogenous tissue flap reconstruction including: pedicled and/or free TRAM flap or DIEP flap reconstruction
* Patients at least 21 years of age
* Patients at least 1 year from the time of mastectomy or completion of immediate, postmastectomy reconstruction

Exclusion Criteria:

Patients who have had any of the following:

* delayed reconstruction (no reconstruction immediately after mastectomy)
* combined autogenous tissue/implant breast reconstruction
* tissue expander
* Patients who have a history of complex regional pain syndrome
* implant explantation (device is removed prematurely due to complications)

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited by their attending surgeon when they return to their surgeon's office for a postoperative appointment following their qualifying surgery
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2006-06; Primary Completion 2021-04-07 (Actual); Study Completion 2021-04-07 (Actual)

PRIMARY OUTCOMES:
Evaluate the degree of touch, vibration, superficial pain, and temperature sensation recovered in the postmastectomy as well as in the reconstructed breast and to compare the sensations recovered in the different groups. | 1 year

SECONDARY OUTCOMES:
The secondary objective is to compare the sensations recovered following tissue expander/implant breast reconstruction with sensations recovered following autogenous tissue reconstruction. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Babak Mehrara, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering web site — http://www.mskcc.org